CLINICAL TRIAL: NCT02176928
Title: Sleep-Disordered Breathing in Chronic SCI: A Randomized Controlled Trial of Treatment Impact on Cognition, Quality of Life, and Cardiovascular Disease
Brief Title: Sleep-Disordered Breathing in Chronic SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Wayne State University (Other)
Responsible Party: Principal Investigator, Shirin Shafazand, Associate Professor of Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20130161; # W81XWH-13-1-0479 (Other Grant/Funding Number: Department of Defense (DoD))
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injury; Sleep Apnea, Obstructive
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AutoPAP (Active Comparator): PAP treatment will be delivered for four months by an auto-titrating device (IntelliPAP AutoAdjust®). These devices automatically set the level of delivered pressure to ensure upper airway patency, to treat detected apneas and hypopneas.
  Interventions: Device: AutoPAP
- Sham PAP (Sham Comparator): Sham PAP treatment will be delivered for four months by an auto-PAP device (IntelliPAP AutoAdjust®) that is set to a fixed low pressure of 3 cmH20 without an ability to titrate according to detected respiratory events.
  Interventions: Device: Sham PAP

INTERVENTIONS:
Device: AutoPAP — PAP will be delivered by an auto-titrating device (IntelliPAP AutoAdjust®). These devices automatically set the level of delivered pressure to ensure upper airway patency, to treat detected apneas and hypopneas.
  AutoPAP treatment 7 nights a week for four months (16 weeks).
  Other Names: IntelliPAP AutoAdjust®; CPAP
  Arms: AutoPAP
Device: Sham PAP — Sham PAP treatment will be delivered by an auto-PAP device (IntelliPAP AutoAdjust®) that is set to a fixed low pressure of 3 cmH20 without an ability to titrate according to detected respiratory events. The pressure is too low to eliminate respiratory events and serves as sham or sub-therapeutic PAP.
  Sham PAP treatment 7 nights a week for four months (16 weeks)./
  Arms: Sham PAP

SUMMARY:
The purpose of this study is to examine impact of Sleep Disordered Breathing (SDB) treatment in persons with chronic Spinal Cord Injury (SCI). The central hypothesis is that the treatment of SDB with Positive Airway Pressure (PAP) will improve cognition, sleep quality, health related quality of life (HRQOL), pain and Cardiovascular Disease (CVD) surrogate measures in persons with chronic SCI.

DETAILED DESCRIPTION:
Investigators will examine the effect of PAP therapy and sleep apnea on thinking (especially memory, learning and concentration), sleep quality, and risks for future heart (cardiovascular) problems in persons with chronic spinal cord injury (SCI).

SDB is a condition where there are pauses in breathing or shallow breathing during sleep due to airway narrowing. This leads to low oxygen levels during sleep and sleep disruption. The usual treatment for sleep apnea is PAP (Positive Airway Pressure) worn while sleeping. This involves the use of usually a mask connected to a machine that supplies enough pressure to keep the airway open during sleep.

SDB will be diagnosed in SCI participants using unattended portable level II polysomnography (PSG) (a portable at home sleep study for one night).

Sleep quality (SQ), SDB risk, insomnia severity, daytime sleepiness,and mood will be measured using questionnaires.

Cognitive evaluations will be completed prior to randomization on all participants who also complete a portable PSG to evaluate general and pre-morbid function, immediate verbal memory, simple and sustained attention, processing speed, and executive function.

Blood and urine samples will be taken for participants with SDB diagnosis after randomization.

All randomized subjects will be fitted with a nasal or full-face mask and head gear. PAP will be delivered by an auto-titrating device. These devices automatically set the level of delivered pressure to ensure upper airway patency, to treat detected apneas, and hypopneas. All subjects will be instructed to use the device nightly during sleep, for the ensuing four months. All outcome measurements will be reassessed after four months of PAP.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tetraplegia or paraplegia (C4-L1)
* American Spinal Injury Association (ASIA) Impairment Scale A, B, C or D
* 18 years and older
* At least one year post injury
* Hearing and vision suitable for comprehension of instructions, and perception of cognitive test stimuli
* No color blindness as measured by a brief screen with color perception Ishihara cards
* Stable medical condition for 2 weeks prior to enrollment. Patients admitted to hospital will be eligible for enrolment if the acute illness precipitating admission is in recovery phase for 2 weeks or longer

Exclusion Criteria:

* Diagnosis of SDB and successful positive airway pressure (PAP) therapy prior to injury. Those with a diagnosis of SDB post injury who are not receiving therapy for SDB (PAP, surgical, and/or oral appliance) are eligible for study enrollment
* Patients who are intubated, have a tracheostomy, and/or are using long term invasive/non-invasive positive pressure ventilation
* Participants with predominant central sleep apnea on PSG requiring bi-level PAP therapy
* Severe traumatic brain injury (GCS < 8 at first assessment)
* Unable to understand or read English at a grade 5 level
* Inability to provide informed consent
* Evidence of advanced neurological or systemic disease that may affect cognitive functioning (e.g., Alzheimer's disease, Dementia, Parkinson's disease)
* Significant aphasia or language impairments
* Positive airway pressure therapy may be contraindicated in some patients with the following preexisting conditions:
* severe bullous lung disease
* pneumothorax
* pathologically low blood pressure
* dehydration
* cerebrospinal fluid leak, recent cranial surgery, or trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Shafazand, MD, MS, Principal Investigator — University of Miami Miller School of Medicine; Pulmonary and Critical Care Medicine
Locations (4):
- United States (4):
  - Miami VA Hospital, Miami, Florida
  - Miami Project to Cure Paralysis, University of Miami Miller School of Medicine, Miami, Florida
  - John D Dingell VA Medical Center, Detroit, Michigan
  - Wayne State University, Detroit, Michigan

REFERENCES:
- [Derived] Graco M, Schembri R, Cross S, Thiyagarajan C, Shafazand S, Ayas NT, Nash MS, Vu VH, Ruehland WR, Chai-Coetzer CL, Rochford P, Churchward T, Green SE, Berlowitz DJ. Diagnostic accuracy of a two-stage model for detecting obstructive sleep apnoea in chronic tetraplegia. Thorax. 2018 Sep;73(9):864-871. doi: 10.1136/thoraxjnl-2017-211131. Epub 2018 May 7. PMID 29735608

RESULTS

PARTICIPANT FLOW:
Groups:
- AutoPAP: PAP treatment will be delivered for four months by an auto-titrating device (IntelliPAP AutoAdjust®). These devices automatically set the level of delivered pressure to ensure upper airway patency, to treat detected apneas and hypopneas.
  AutoPAP: PAP will be delivered by an auto-titrating device (IntelliPAP AutoAdjust®). These devices automatically set the level of delivered pressure to ensure upper airway patency, to treat detected apneas and hypopneas.
  AutoPAP treatment 7 nights a week for four months (16 weeks).
- Sham PAP: Sham PAP treatment will be delivered for four months by an auto-PAP device (IntelliPAP AutoAdjust®) that is set to a fixed low pressure of 3 cmH20 without an ability to titrate according to detected respiratory events.
  Sham PAP: Sham PAP treatment will be delivered by an auto-PAP device (IntelliPAP AutoAdjust®) that is set to a fixed low pressure of 3 cmH20 without an ability to titrate according to detected respiratory events. The pressure is too low to eliminate respiratory events and serves as sham or sub-therapeutic PAP.
  Sham PAP treatment 7 nights a week for four months (16 weeks)./
Period: Overall Study
Arm/Group | AutoPAP | Sham PAP
Started | 21 | 21
Completed | 19 | 17
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AutoPAP | Sham PAP | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.6) | 46.9 (14.3) | 44.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 6 | 23
  Not Hispanic or Latino | 4 | 14 | 18
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 16 | 13 | 29
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Functioning as Measured by PASAT
Description: Paced Serial Addition Test (PASAT) measures divided attention and memory. PASAT has a total score ranging from 0 to 60 with the lower scores indicate greater impairment of attention.
Time Frame: 16 weeks
Population: 2 sham participants did not complete PASAT at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AutoPAP | Sham PAP
Number analyzed (Participants) | 19 | 15
score on a scale | 10.6 (7.6) | 15.2 (10.4)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | AutoPAP | Sham PAP
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
only 39% of subjects were using PAP more than 4 hours a night by end of week 1 and this number dropped to less than 30% by end of month 4, this may impact final conclusions. Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT02176928/Prot_SAP_000.pdf